CLINICAL TRIAL: NCT04346407
Title: Impact of Dronabinol on Post-operative Pain After Lumbar Fusion for Degenerative Disorders of the Spine
Brief Title: Dronabinol for Post-operative Pain After Lumbar Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jeffrey L Gum MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey L Gum MD, Attending Spine Surgeon, Norton Leatherman Spine Center
Organization: Norton Leatherman Spine Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20.N0042
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Post-operative Pain
Keywords: Lumbar Fusion; Post-operative Opioid Consumption; Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dronabinol; Capsules

STUDY DESIGN:
Intervention Model Description: Double-blind Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo, randomization and blinding will be maintained by the Hospital Pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronabinol (Experimental): 2.5mg of oral Dronabinol daily starting with pre-op cocktail and continued twice daily for three days after surgery
  Interventions: Drug: Dronabinol 2.5mg Cap
- Placebo (Placebo Comparator): Capsule with placebo daily starting with pre-op cocktail and continued twice daily for three days after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 2.5mg Cap — 2.5mg of oral Dronabinol daily starting with pre-op cocktail and continued twice daily for three days after surgery
  Other Names: Marinol; Syndros
  Arms: Dronabinol
Drug: Placebo — Placebo capsule daily starting with pre-op cocktail and continued twice daily for three days after surgery
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
Impact of 2.5mg of oral Dronabinol daily versus placebo on post-operative opioid consumption on patients aged 18 to 65 years old undergoing 1 to 3 level posterolateral fusion

DETAILED DESCRIPTION:
This is a randomized double-blind clinical trial comparing 2.5mg of oral Dronabinol daily starting with pre-op cocktail and continued twice daily for three days after surgery versus placebo for patients aged 18 to 65 years old undergoing 1 to 3 level posterolateral fusion. The outcome of interest is post-operative opioid consumption defined as cumulative Morphine Milligram Equivalents at 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old
* Patients undergoing 1 to 3 level posterolateral fusion
* Opioid naïve or not
* No prior spine fusion
* Willing and able to sign an Informed Consent

Exclusion Criteria:

* Indication for surgery is fracture, tumor or infection
* Comorbid psychiatric diagnosis requiring therapy and/or medication
* Comorbid chronic pain syndrome (reflex sympathetic dystrophy, fibromyalgia)
* Has hepatic disease
* On workers compensation/disability/litigation
* Known adverse reaction to medications to be administered
* History of alcohol and drug abuse
* On long-acting narcotic pain medication (including extended release narcotic pain medications and methadone)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative Morphine Milligrams at 72 hours post-operative | 72 hours post-operative
  Cumulative Morphine Milligrams consumed in-hospital 72 hours after surgery

SECONDARY OUTCOMES:
Cumulative Morphine Milligrams at 24 hours post-operative | 24 hours post-operative
  Cumulative Morphine Milligrams consumed in-hospital 24 hours after surgery
Cumulative Morphine Milligrams at 48 hours post-operative | 48 hours post-operative
  Cumulative Morphine Milligrams consumed in-hospital 48 hours after surgery
Worst pain in past 24 hours post-operative | 24 hours post-operative
  Worst pain in past 24 hours post-op on a scale of 0 to 10, with 0 as no pain and 10 as worst pain imaginable
Worst pain in past 48 hours post-operative | 48 hours post-operative
  Worst pain in past 48 hours post-op on a scale of 0 to 10, with 0 as no pain and 10 as worst pain imaginable
Worst pain in past 72 hours post-operative | 72 hours post-operative
  Worst pain in past 72 hours post-op on a scale of 0 to 10, with 0 as no pain and 10 as worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Gum, MD, Principal Investigator — Norton Healthcare
Locations (1):
- Norton Healthcare, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No